CLINICAL TRIAL: NCT05065268
Title: Visual Rehabilitation in a Pediatric Population of Patients With Homonymous Hemianopia: a Pilot Study on Virtual-reality Stimulation
Brief Title: Visual Rehabilitation in Children With Homonymous Hemianopia: a Pilot Study on Virtual-reality Stimulation
Acronym: HH-IVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Eric Bouffet, Head of Pediatric Neuro-oncology, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1000076413
Record Dates: First submitted 2021-08-31; First posted 2021-10-04 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Hemianopia; Brain Tumor; Children, Only
Keywords: hemianopia; Brain tumor; children
MeSH Terms: conditions — Hemianopsia; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Visual rehabilitation using home based audiovisual rehabilitation in immersive virtual reality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interventional (Experimental): Immersive virtual-reality stimulation (IVR): 1 session of 3 blocks of 15 trials of 20 seconds each. Rest time is 1-2 minute(s) between blocks. 1 session lasts 19 minutes.1 session every 2 days for 4 weeks (15 sessions total).
  Interventions: Device: Immersive Virtual-Reality Stimulation

INTERVENTIONS:
Device: Immersive Virtual-Reality Stimulation — IVR stimulation every 2 days (± 1 day) at any time during the day (delivery).

SUMMARY:
There are currently no visual rehabilitation strategies for children presenting visual field defects consecutive to a brain tumor or its treatment. This study seeks to investigate the use of a home-based stimulation visual rehabilitation program using immerse-virtual reality (IVR) in children aged 4-10 years old with a diagnosis of hemianopia

DETAILED DESCRIPTION:
A brain tumor and its treatment can affect the visual system at different levels, from the optic nerves (through compression or infiltration). Children with brain tumors can present visual impairments like decreased visual acuity and contrast sensitivity, loss of color vision, and visual field loss such as hemianopias. Patients with hemianopia present difficulties in detecting stimuli in the defective visual field and show defective scanning and exploration. Moreover, they show a rotation and compression of the auditory space leading to imprecise localization of sound across both hemispaces. Patients with hemianopia naturally develop oculomotor strategies to compensate for visual field loss, but visual rehabilitation procedures must still be developed to optimize/improve visual perception in the blind field. Several studies demonstrated that these patients could improve visual perception in the damaged hemifield after a stimulation procedure where auditory and visual stimuli were temporally and spatially correlated. Such audiovisual stimulation programs induce a functional and anatomical reorganization of the visual connectivity in subcortical and cortical structures over time.

The current strategies rely on a significant workload, over 30 hours of audiovisual stimulation using static, spatially, and temporally coherent stimuli displayed on large screens/panels in a clinical setting. These strategies require frequent visits to the clinic impeding the patients' adherence and compliance and increasing the burden of disease. We seek to develop an audiovisual stimulation procedure using immersive virtual reality (IVR) using a head-mounted display (HMD). This is an emerging and very promising visual rehabilitation approach using high-technology devices. It is developed to provide sensory stimulation with better ecological validity due to virtual reality, greater flexibility due to home-based programs, and improved efficiency due to patient-tailored protocols. IVR is a versatile technology, allowing its potential use for the rehabilitation of a variety of low-vision conditions. There are currently limited practical results on whether this technology is suitable for low-vision patients to use at home and if it can be deployed on a large scale. A few case reports/series studies suggested the potential effectiveness of IVR on visual perception in teenagers, adults, and the elderly but more information as to the potential of use and effectiveness of this technology in children and young teenagers is necessary

ELIGIBILITY:
Inclusion Criteria:

1. Homonymous hemianopsia
2. Male and female.
3. > 8 years old
4. Interpupillary distance >=56 mm
5. BCVA > 20/200
6. Ability to follow visual and auditory stimuli and training instructions.
7. Home Wi-Fi access.

Exclusion Criteria:

1. Ocular diseases
2. Both eyes with media opacity that impairs microperimetry testing.
3. Inability to perform during testing and training.
4. Consumption of psychoactive drugs.
5. 3 consecutive VRISE scores < 25 at inclusion.
6. History of vertigo or dizziness
7. Prior vision rehabilitation interventions.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Feasibility and effectiveness of a home based audiovisual stimuaton in immersive virtual-reality to restore visual perception in children with brain tumour associated hemianopia. | 7 months
  Feasibility objectives for our pilot study to be considered successful
  1. . Number of patients completing the stimulation protocol: ≥ 8 out of 10 patients (80%).
  2. . Number of IVR sessions performed by the patients to consider the stimulation protocol complete: ≥ 12 sessions out of 15 (80%).
  3. . Number of consecutive virtual-reality induced symptoms and effects (VRISE) scores < 25: ≤ 3 per patient during the treatment period.
  4. . Number of patient drop-outs due to cybersickness (discomfort symptoms experienced in VR): ≤ 2 (20%) during the treatment period.

SECONDARY OUTCOMES:
Change in Visual acuity | 7 months
  Corresponds to the potential effectiveness of IVR stimulation in visual acuity assessed by standard procedures by ophthalmologists.
  -Best Corrected Visual Acuity, distance, and near vision (range 20/12.5 to <20/1000, higher score = better outcome)
Change in Reading speed | 4 weeks
  This corresponds to the potential effectiveness of IVR stimulation in reading speed assessed by standard procedures by ophthalmologists.
  Endpoints will measure change from baseline at 2 and 4 weeks in:
  -Mean reading speed (Minnesota Low Vision Reading test, MNREAD - range 0 words/minute to 280 words/minute, higher score = better outcome)
Change in Field of vision | 4 weeks
  This corresponds to the potential effectiveness of IVR stimulation in the field of vision assessed by standard procedures by ophthalmologists.
  Endpoints will measure change from baseline at 2 and 4 weeks in:
  -Mean contrast sensitivity (Functional Acuity Contrast Test, FACT - range 0.48 cyc./deg. to 2.41 cyc./deg., higher score = better outcome)
Change in Quality of life | 4 weeks
  This corresponds to the potential effectiveness of IVR stimulation in the quality of life.
  Endpoints will measure change from baseline at 2 and 4 weeks in:
  -Quality of life scores (Children's Vision Function Questionnaire, higher score = better outcome).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - The Hospital for Sick Children, Toronto, Ontario
  - University Health Network, Toronto, Ontario

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05065268/Prot_SAP_000.pdf